CLINICAL TRIAL: NCT00059046
Title: Kinetic Studies in Whole Body and Brain of [11C]DASB PET Imaging of Serotonin Transporters
Brief Title: Brain Imaging of Serotonin Transporters in the Brain
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030159; 03-M-0159
Record Dates: First submitted 2003-04-16; First posted 2003-04-16 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Healthy; Serotonin Transporter
Keywords: Neuroreceptors; PET Measurements; Kinetic Analysis; Test/Retest; Healthy Volunteer; HV

SUMMARY:
Serotonin is a chemical involved in the regulation of emotions, anxiety, sleep, stress, and other body functions. The purpose of this study is to use brain imaging technology to study how serotonin works in the brain.

The serotonin transporter (SERT) regulates the release of sertonin throughout the body. Until recently, radioactive chemicals called tracers were not suitable for viewing SERT activity. However, a newly developed tracer called [11C]DASB can be used with positron emission tomography (PET) imaging to view the parts of the brain that use serotonin.

Participants in this study will be screened with medical and psychiatric examinations, an electrocardiogram (EKG), and blood and urine tests. This study comprises two parts. During Part 1, participants will undergo a whole-body PET scan. During Part 2, participants will undergo a magnetic resonance imaging (MRI) scan of the brain. At the next study visit, participants will have one or two PET head scans. If not is not possible to perform both scans on the same day, an additional visit will be scheduled for the second PET scan.

DETAILED DESCRIPTION:
The serotonin transporter (SERT) modulates the activity of the central serotonergic system and SERT is also the primary target of the widely prescribed specific serotonin reuptake inhibitors. Until recently, suitable radioligands for in vivo imaging of SERT have not been available. However, a recently developed PET radioligand, [11C]DASB, appears suitable for quantifying SERT in humans. In the two protocols that have been approved by the CSRP for submission to the IRB, we planned to use [11C]DASB PET to study the pathophysiology of SERT in Parkinson's disease and OCD. This protocol was created to address criticisms raised by the NIH RDRC committee and the external scientific review.

1. The NIH RDRC (Radioactive Drug Research Committee) review of this protocol asked that we obtain human biodistribution data to confirm the expected low levels of radiation exposure, based upon our prior studies in monkeys.
2. To address one of the criticisms raised by the CSRP review, namely 1) to quantify SERT binding parameters with [11C]DASB in up to 10 normal subjects and 2) to determine the reliability and reproducibility of SERT binding parameter measurements by performing a second retest [11C]DASB PET study in the same subjects, because such data are not available for this radioligand. PET scanning will be performed with an intravenous injection of 20 mCi of [11C]DASB for 2 h, during which multiple arterial blood samples will also be obtained. The reproducibility of SERT binding parameters will be assessed by calculating the variability as well as the intraclass correlation coefficient between test/retest measurements. We expect that 1) we can accurately quantify SERT binding parameters using [11C]DASB PET imaging and 2) [11C]DASB PET measurements of SERT binding will be reliable and reproducible.

ELIGIBILITY:
INCLUSION CRITERIA: WHOLE BODY IMAGING

Diagnosis: Healthy

Ages: 18-50 years

EXCLUSION CRITERIA: WHOLE BODY IMAGING

History of psychiatric disease, substance dependence or traumatic brain injury, severe systemic disease, poor vision or hearing.

History of substance abuse within 6 months

Abnormal laboratory tests, including HIV test

Any prior participation in other research protocols involving radiation exposure within the past year

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits

Pregnancy and Breast Feeding

Positive HIV test

INCLUSION CRITERIA: PART 2 KINETIC

Age: 18-50 y

Male or female

Consent given

EXCLUSION CRITERIA: PART 2 KINETIC

DSM-IV Axis I diagnostic criteria such as history of, or current diagnosis ADHD, mood/anxiety disorder, alcohol or psychoactive substance abuse/dependence. All subjects must meet none of the Axis I diagnoses.

Psychotropic medication or other drugs that may cross the blood brain barrier. Drug free period must be greater than 4 weeks (antidepressants and benzodiazepine) and greater than 6 weeks (fluoxetine, antipsychotics, anticonvulsants).

Pregnancy or breastfeeding

Abnormal MRI other than minor atrophy

Abnormal laboratory tests, including HIV test

Claustrophobia

Pregnancy or breast feeding. Women with child bearing potential will a pregnancy test to exclude pregnancy

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits. Limits: A total effective dose or 5.0 rem in a year.

Any condition that increases risk for MRI (e.g., pacemaker, metallic foreign body in the eye, etc.)

Traumatic brain injury, severe systemic disease, poor vision or hearing

Major medical conditions or neurological disorders

Single radial and ulnar arterial circulation. This will be determined during physical examination (A simple wrist compression test)

Individuals who recently donated blood.

Unable to lay on one's back for PET/MRI scans. PET and MRI scans take approximately 2 and 1 hours, respectively.

Novacaine allergy - yes - Local anesthetic used for insertion of arterial and venous catheters.

Positive HIV test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2003-04; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cash R, Raisman R, Ploska A, Agid Y. High and low affinity [3H]imipramine binding sites in control and parkinsonian brains. Eur J Pharmacol. 1985 Oct 29;117(1):71-80. doi: 10.1016/0014-2999(85)90473-x. PMID 3002804
- [Background] Raisman R, Cash R, Agid Y. Parkinson's disease: decreased density of 3H-imipramine and 3H-paroxetine binding sites in putamen. Neurology. 1986 Apr;36(4):556-60. doi: 10.1212/wnl.36.4.556. PMID 2938025
- [Background] Crow TJ, Cross AJ, Cooper SJ, Deakin JF, Ferrier IN, Johnson JA, Joseph MH, Owen F, Poulter M, Lofthouse R, et al. Neurotransmitter receptors and monoamine metabolites in the brains of patients with Alzheimer-type dementia and depression, and suicides. Neuropharmacology. 1984 Dec;23(12B):1561-9. doi: 10.1016/0028-3908(84)90100-x. PMID 6084823